CLINICAL TRIAL: NCT07361952
Title: Oral Versus Intravenous Fluid Therapy in the Emergency Department
Acronym: OVID-B
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Esbjerg Hospital - University Hospital of Southern Denmark (Other)
Collaborators: Odense University Hospital (Other); Hospital of Southern Jutland, Aabenraa, Denmark (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S-20250042
Record Dates: First submitted 2025-12-29; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Fluid Management
Keywords: oral fluids; Emergency department; intravenous fluids; fluid management
MeSH Terms: conditions — Emergencies | interventions — Fluid Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravenous fluids (Active Comparator): Participants randomized to receive IV crystalloid fluids during ED stay
  Interventions: Other: Intravenous fluids
- Oral fluids (Experimental): Participants randomized to receive oral tap water during ED stay
  Interventions: Other: Oral fluids

INTERVENTIONS:
Other: Oral fluids — Any fluid volume prescribed by the physician during the ED stay is administered orally.
  Arms: Oral fluids
Other: Intravenous fluids — Any fluid volume prescribed by the physician during the ED stay is administered intravenously.
  Arms: Intravenous fluids

SUMMARY:
The goal of this randomized clinical feasibility trial is to determine whether oral fluid therapy can achieve prescribed fluid volumes as effectively as intravenous fluid therapy in adult patients admitted to the emergency department who require fluid treatment.

The main questions it aims to answer are:

Are patients receiving oral fluids equally likely to achieve the prescribed fluid volume compared with patients receiving intravenous fluids?

Is it feasible to conduct a randomized trial of oral versus intravenous fluid therapy in the emergency department, based on recruitment rate and protocol adherence?

Researchers will compare oral tap water administration with standard intravenous crystalloid therapy to assess whether oral fluids are non-inferior in achieving prescribed fluid volumes and to evaluate feasibility outcomes.

Participants will:

Be randomized to receive either oral tap water or intravenous crystalloid fluids during their stay in the emergency department

Receive a fluid volume and administration rate determined by the treating physician

Be monitored according to standard clinical practice during the emergency department stay

Have fluid intake, vital signs, and clinical outcomes recorded, with follow-up through routine health records up to 30 days after inclusion

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or above
* At least 1000 ml of crystalloid fluid therapy prescribed by the physician

Exclusion Criteria:

* Altered mental state prohibiting oral fluid intake (Glasgow Coma Scale ≤ 12)
* Pregnancy
* Oral fluids contraindicated (e.g. bowel obstruction)
* Severe hyponatremia (sodium <120 mEq/L)
* Requiring treatment in the intensive care unit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-10-03 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients achieving the fluid volume prescribed during the first 48 hours in the emergency department | From inclusion until end of participation. End of participation is defined as the timepoint of leaving the emergency department or after 48 hours, whichever happens first.

SECONDARY OUTCOMES:
Fluids received in the ED (ml) | From inclusion to end of participation (defined as ED stay or maximum of 48 hours), unless mentioned otherwise
  Intravenous fluids, oral fluids, total fluids
Fluids received in the ED after inclusion in the study (ml) | From inclusion to end of participation (defined as ED stay or maximum of 48 hours), unless mentioned otherwise
  Intravenous fluids, oral fluids, total fluids
Change in systolic and mean arterial pressure at 8 hours or discharge, whatever comes first. | 8 hours or discharge, whatever comes first.
Hospital-free days alive at 30 days (counting up to the day the patient deceased if applicable) | 30 days
Mortality at 30 days | 30 days
Number of hours with a peripheral intravenous catheter | From inclusion to end of participation (defined as ED stay or maximum of 48 hours), unless mentioned otherwise

CONTACTS AND LOCATIONS:
Locations (3):
- Denmark (3):
  - Emergency Department, South Jutland Hospital, Aabenraa
  - Emergency Department, Esbjerg Hospital, Esbjerg
  - Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD available upon reasonable request, subject to approval and data protection regulations.
Supporting Information: Study Protocol
Time Frame: Data will be available upon reasonable request beginning after publication of the primary results and ending 5 years thereafter.
Access Criteria: Access to de-identified individual participant data (IPD) and supporting documentation will be granted to qualified researchers upon reasonable request. Requests must include a written proposal describing the research question, planned analyses, and intended use of the data. Proposed analyses must be scientifically sound and consistent with the scope of the original study.
  Requests will be reviewed by the study investigators to assess scientific merit, feasibility, and compliance with ethical approvals and data protection regulations. Where required, approval from relevant ethics committees or data protection authorities must be obtained prior to data access.
  Data sharing will be subject to the execution of a data sharing agreement outlining the terms of use, data security requirements, and restrictions on onward sharing. Data will be provided in a secure format and access will be limited to the approved analyses.